CLINICAL TRIAL: NCT03159832
Title: Safety and Pharmacokinetics/Pharmacodynamics of SHR3824 in Type 2 Diabetes Patients With Renal Insufficient (Open-label, Parallel-Group, Single-Dose Study)
Brief Title: Safety and Pharmacokinetics/Pharmacodynamics of SHR3824 in Type 2 Diabetes Patients With Renal Insufficient
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR3824-110
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2016-06

CONDITIONS: Renal Insufficiency,Type 2 Diabetes
Keywords: Efficacy; PK/PD study; Renal Insufficiency; Type 2 Diabetes
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus, Type 2 | interventions — henagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal renal function (Active Comparator): All subjects were given SHR3824 20mg only one time.
  Interventions: Drug: SHR3824
- Mild renal dysfunction (Active Comparator): All subjects were given SHR3824 20mg only one time.
  Interventions: Drug: SHR3824
- Moderate renal dysfunction (Active Comparator): All subjects were given SHR3824 20mg only one time.
  Interventions: Drug: SHR3824

INTERVENTIONS:
Drug: SHR3824 — All subjects were given SHR3824 20mg only one time.

SUMMARY:
The purpose of the study is to investigate the pharmacokinetics/pharmacodynamics and safety of SHR3824 in Type 2 Diabetes Patients with Renal Insufficient.

DETAILED DESCRIPTION:
This trial was a parallel, open-label, single dose study. The subject was divided into one of three groups according to the degree of renal Insufficiency,including normal, mild and moderate. All subjects were given SHR3824 20mg, the blood and urine samples were collected before and after dosing.

ELIGIBILITY:
Inclusion Criteria:

* with a body mass index(BMI) between 19 and 33 Kg/m2;
* The estimated glomerular filtration rate (eGFR)of subjects in groups must meet the corresponding standards:mild renal insufficiency:60 to 89 ml/min/1.73m2;Moderate renal insufficiency: 30 to 59 ml/min/1.73m2.
* Had signed the informed consent himself or herself voluntarily.

Exclusion Criteria:

* Urinary tract infections, or vulvovaginal mycotic infections
* Suspected or diagnosed as kidney cancer or other malignancies in patients
* Autoimmune kidney disease, history of renal transplantation, dialysis patients being treated
* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to SHR3824,SGLT2 inhibitor analogs, or any other structural analogs
* Alcohol, tobacco, drug abusers;alcohol abuse is defined as a day for regular alcohol consumption more than the following standards: beer 570 ml, light beer 750 ml, red wine 200 ml, white wine 60 ml, which including about 20g alcohol;Tobacco is defined as five or more per day.
* Pregnancy or lactation women, or a fertility male or female is not willing to contraception during test.
* Researchers considered that there was any situation that may cause the participants can't finish this study or bring any obvious risk to subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve (AUC) of SHR3824 | 72 hours after dosing
  AUC (a measure of the body's exposure to SHR3824) will be compared between normal renal function patients and mild or moderate renal dysfunction patients
The maximum plasma concentration (Cmax) of SHR3824 | 72 hours after dosing
  Cmax (a measure of the body's exposure to SHR3824) will be compared between normal renal function patients and mild or moderate renal dysfunction patients

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | 72 hours after dosing
  The number of volunteers with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese people's liberation army general hospital of Chengdu military area, Chengdu, Sichuan, China